CLINICAL TRIAL: NCT03409263
Title: Österreichisches Register (inklusive Biobank) Für Transjuguläre Intrahepatische Portosystemischem Shunts (TIPS): AUTIPS (AUstrian TIPS Study)
Brief Title: Austrian Registry on Transjugular Intrahepatic Portosystemic Shunts
Acronym: AUTIPS
Status: Recruiting | Type: Observational
Sponsor: Thomas Reiberger (Other)
Collaborators: Austrian Association of Gastroenterology and Hepatology (Other)
Responsible Party: Sponsor-Investigator, Thomas Reiberger, Univ. Prof. Priv.-Doz. Dr., Medical University of Vienna
Organization: Medical University of Vienna (Other)
Other Study IDs: AUTIPS 1943/2017
Record Dates: First submitted 2018-01-18; First posted 2018-01-24 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Portal Hypertension
Keywords: Cirrhosis; Advanced chronic liver disease; Ascites; Variceal hemorrhage; Transjugular intrahepatic portosystemic shunt
MeSH Terms: conditions — Hypertension, Portal; Fibrosis; Ascites | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — Blood samples (collected during routine blood draws): chemistry, hematology, coagulation panel Ascites: WBC, PMN, protein Urine assessment: RBC, protein, sediment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Observational study — Not applicable (observational registry study)

SUMMARY:
Patients with TIPS will be recruited in this prospective registry study. The clinical course will be documented and biomarkers for prediction of complicatiosn will be assessed.

DETAILED DESCRIPTION:
Patients with advanced chronic liver disease may develop portal hypertension, which is the main cause for most complications and deaths of patients with liver cirrhosis. Implantation of a transjugular intrahepatic portosystemic shunt (TIPS) leads to instantaneous alleviation of portal hypertension, but may cause hepatic encephalopathy. Stent grafts, as well as patient stratification and medical surveillance, have drastically improved over the past decades. However, there are few data on long-term outcome after TIPS implantation.This prospective registry study will assess the clinical course of patients after undergoing TIPS intervention and biomarkers for complications after TIPS implantation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-99 years
* Portal hypertension
* Anticipated or past implantation of a transjugular intrahepatic portosystemic shunt (TIPS)
* Informed consent

Exclusion Criteria:

* Retraction of consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients or outpatients who are scheduled for TIPS implantation, or who have recently undergone TIPS implantation and are visiting outpatienc clinics for control visits/surveillance
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2018-03-28 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Transplant-free survival | 0-10 years
  Assessment of transplant-free survival after TIPS implantation

SECONDARY OUTCOMES:
Assessment of portalhypertensive complications | 0-10 years
  Incidence of portalhypertensive complications
Assessment of hepatic encephalopathy | 0-10 years
  Incidence of hepatic encephalopathy
Assessment of Patient Reported Quality of Life (SF36v2) | 0-10 years
  Validated Questionnaire: SF36v2 pre TIPS and after TIPS. The SF36 consists of 36 items measuring 8 domains: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health.
  The mental (MCS) and physical (PCS) component summary scores, as the main read-outs of the SF-36 form, can be regarded as physiological ('normal') when the calculated score lies between 45 and 55, because the results are normalized to a normal "reference" population assigned 50 points. Scores below 45 define worse-than-average physical (PCS) or mental (MCS) health, while scores above 55 indicate better-than-average physical (PCS) or mental (MCS) health, when compared to a normal population.
Assessment of Patient Reported Quality of Life (CLDQ) | 0-10 years
  Validated Questionnaire CLDQ pre TIPS and after TIPS The CLDQ includes 29 items in the following domains: abdominal symptoms, fatigue, systemic symptoms, activity, emotional function and worry. The responses in the 29 CLDQ items, respectively, are recorded on scales ranging from in 1 ("none of the time") to 7 ("all of the time").

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Reiberger, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No
Individual participant data may not be shared publicly due to local data safety regulations. Please contact the sponsor for more information.